CLINICAL TRIAL: NCT03462368
Title: Effects of Photobiomodulation and Antimicrobial Photodynamic Therapy Associated With Subepithelial Connective Tissue Graft on the Root Coverage of Multiple Gingival Recessions: A Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Root Coverage by Connective Graft and Different Root Conditioning Adjunctive Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOBaPDTrecession
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Gingival Recession; Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession | interventions — Tooth Exfoliation; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Root surface treatment by scaling and root planing
  Interventions: Procedure: Control
- antimicrobial photodynamic therapy (Experimental): Root surface treatment by antimicrobial photodynamic therapy
  Interventions: Procedure: antimicrobial photodynamic therapy
- Photobiomodulation (Active Comparator): Treatment of the whole surgical site with laser
  Interventions: Procedure: Photobiomodulation

INTERVENTIONS:
Procedure: Control — In the procedure of subepithelial connective tissue graft, exposed dental roots will be treated by scaling and root planing only.
  Other Names: Scaling and root planing only
  Arms: Control
Procedure: antimicrobial photodynamic therapy — In the procedure of subepithelial connective tissue graft, exposed dental roots will be treated by antimicrobial photodynamic therapy with toluidine blue O (10mg/ml)
  Arms: antimicrobial photodynamic therapy
Procedure: Photobiomodulation — After the procedure of subepithelial connective tissue graft the whole surgical site will receive red laser application.
  Other Names: Low level laser therapy
  Arms: Photobiomodulation

SUMMARY:
The aim of this study was to evaluate the effect of two different treatment agents used in conjunction with subepithelial connective graft technique on root coverage outcomes in multiple recession defects. Half of patients will receive root treatment with antimicrobial photodynamic therapy and the other half will receive photobiomodulation therapy by laser on surgery site.

DETAILED DESCRIPTION:
Antimicrobial photodynamic therapy has been widely used in Periodontics to obtain reduction of periodontopathogenic bacteria with absence of systemic side effects and minimal bacterial resistance. Also, it has properties of root demineralization and exposure of collagen fibers. These properties may enhance root coverage in procedures of subepithelial connective graft. Laser photobiomodulation has the potential to increase healing and repair, this can generate gains in the root coverage and dental hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Gingival recession - two or more Miller's class I or II (2 to 5 mm of height)
* Indication of root coverage by dentin hypersensitivity or esthetic.
* Minimum palate thickness (1,5mm)
* Visible Enamel cement junction (JCE) on the teeth to be treated and pulp vitality
* Patients without signs of periodontal disease activity and with plaque index and bleeding on probing throughout ≤20%;

Exclusion Criteria:

* Use of drugs that affect periodontal tissues (eg: anticonvulsants, calcium channel blockers, cyclosporine, bisphosphonates, hormone-based contraceptives, steroids)
* Smokers
* Pregnancy
* Diabetics
* History of head and neck radiotherapy
* Teeth with mobility
* Malpositioned teeth
* History of periodontal surgery at the area on the last 12 months
* Patients with orthodontic therapy in progression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Total root coverage | One year
  Total root coverage measured with a periodontal probe in millimeters. Ideal if the distance from cemento-enamel junction to gingival margin = 0 mm

SECONDARY OUTCOMES:
Keratinized mucosa width | One year
  Keratinized mucosa width is measured with a periodontal probe in mm, from gingival margin to mucogingival junction. Ideal if keratinized mucosa width > 5mm
Probing depth | One year
  Probing depth measured with a periodontal probe in millimeters. The distance from gingival margin and the apical point of gingival pocket or sulcus. Ideal if <2mm.
Clinical attachment level | One year
  Clinical attachment level measured with a periodontal probe in millimeters. The distance from cemento-enamel junction and the apical point of gingival pocket or sulcus. Ideal if <2mm.
Dentin hypersensitivity | One year
  Dentin hypersensitivity measured by applying an air jet on teeth and patient fills up a visual analogue scale. Ideal if = 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karam PS, Sant'Ana AC, de Rezende ML, Greghi SL, Damante CA, Zangrando MS. Root surface modifiers and subepithelial connective tissue graft for treatment of gingival recessions: a systematic review. J Periodontal Res. 2016 Apr;51(2):175-85. doi: 10.1111/jre.12296. Epub 2015 Jun 11. PMID 26095265
- [Background] Fernandes-Dias SB, de Marco AC, Santamaria M Jr, Kerbauy WD, Jardini MA, Santamaria MP. Connective tissue graft associated or not with low laser therapy to treat gingival recession: randomized clinical trial. J Clin Periodontol. 2015 Jan;42(1):54-61. doi: 10.1111/jcpe.12328. Epub 2014 Dec 17. PMID 25363203
- [Background] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681
- [Derived] Cardoso MV, Sant'Ana ACP, Zangrando MSR, Damante CA. Effects of photobiostimulation and antimicrobial photodynamic therapy associated with gingival grafts for root coverage: three-arm randomized clinical trial. Lasers Med Sci. 2025 Apr 14;40(1):190. doi: 10.1007/s10103-025-04449-0. PMID 40227516